CLINICAL TRIAL: NCT01800656
Title: Endoloop-assisted Colorectal Polypectomy or "Ligate and Let go" in Patients With Long-term Antiplatelet Therapy
Brief Title: Assessing Endoloop-assisted Polypectomy in Patients With Antiplatelet Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Milutin Bulajic (Other)
Responsible Party: Sponsor-Investigator, Dr Milutin Bulajic, Principal investigator, Hospital Danilo I Cetinje
Organization: Hospital Danilo I Cetinje (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDL-001
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ligate and let go (Experimental): Subjects are submitted to endoloop-assisted "ligate and let go" colorectal polypectomy.
  Interventions: Procedure: Endoloop-assisted "ligate and let go" colorectal polypectomy
- Snare polypectomy (Active Comparator): Subjects are submitted to endoloop-assisted snare colorectal polypectomy
  Interventions: Procedure: Endoloop-assisted snare colorectal polypectomy

INTERVENTIONS:
Procedure: Endoloop-assisted "ligate and let go" colorectal polypectomy — The technique implies placement of endoloop snare on the base of large pedunculated colorectal polyps without consecutive snare polypectomy.
  Arms: Ligate and let go
Procedure: Endoloop-assisted snare colorectal polypectomy — The technique implies placement of endoloop snare on the base of large pedunculated colorectal polyps with consecutive snare polypectomy.
  Arms: Snare polypectomy

SUMMARY:
The aims of this study were to examine: 1) safety and feasibility of antiplatelet therapy interruption 7 days prior to polypectomy in patients with long-term antiplatelet therapy; 2) safety and feasibility of endoloop assisted snare polypectomy in patients with long-term antiplatelet therapy; 3) safety and feasibility of so called "ligate and let go" approach in patients with long-term antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* pedunculated colorectal polyps
* larger than 2cm in diameter
* long-term antiplatelet therapy

Exclusion Criteria:

* presence of intraepithelial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Post-polypectomy bleeding | 24h-15 days

CONTACTS AND LOCATIONS:
Overall Officials: Milutin Bulajic, Dr, Principal Investigator — Hospital Danilo I Cetinje